CLINICAL TRIAL: NCT02772718
Title: An Open-Label Study of XOMA 358 in Patients With Hypoglycemia After Gastric Bypass Surgery
Acronym: XOMA 358
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: XOMA (US) LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X358603
Record Dates: First submitted 2016-05-03; First posted 2016-05-13 (Estimated); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Hypoglycemia
Keywords: Hypoglycemia
MeSH Terms: conditions — Hypoglycemia | interventions — XOMA 358

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 - single dose (Experimental): Cohorts A, B, and C
  Interventions: Drug: XOMA 358 single dose level A; Drug: XOMA 358 single dose level B; Drug: XOMA 358 single dose level C
- Part 2 - multiple doses (Experimental): Cohort 1
  Interventions: Drug: XOMA 358 multiple dose level 1

INTERVENTIONS:
Drug: XOMA 358 single dose level A — XOMA 358 single dose level A administered by intravenous infusion
  Arms: Part 1 - single dose
Drug: XOMA 358 single dose level B — XOMA 358 single dose level B administered by an intravenous infusion
  Arms: Part 1 - single dose
Drug: XOMA 358 single dose level C — XOMA 358 single dose level C administered by an intravenous infusion
  Arms: Part 1 - single dose
Drug: XOMA 358 multiple dose level 1 — XOMA 358 multiple dose level 1 administered by an intravenous infusion
  Arms: Part 2 - multiple doses

SUMMARY:
The purpose of this study is to evaluate the safety and clinical pharmacology of XOMA 358 in patients with hypoglycemia after gastric bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years of age
* Body Mass Index < 35 kg/m2 at baseline, unless discussed with Medical Monitor and patients with higher body mass index do not have significant medical co-morbidities that would confound ability to assess safety and efficacy of study drug.
* Received gastric bypass surgery more than 1 year before dosing
* Occurrence of postprandial hypoglycemia (blood glucose less than 60mg/dL) during the Baseline provocation assessments and/or by continuous glucose monitoring, as defined in the protocol.

Exclusion Criteria:

* History of type 1 diabetes
* Planned use of the following medications on or after Day -3 (Part 1):

  * Any agent for hypoglycemia, such as diazoxide or octreotide
  * Antihyperglycemic agents, including subcutaneous insulin therapy, sulfonylureas, SGLT2 inhibitors, and GLP-1 agonists
  * Systemic glucocorticoids or β agonists that may affect glucose metabolism
  * Long-acting somatostatin analogs or glucose-affecting medications
* During Part 2, the following therapies are prohibited as specified below:

  * Tramadol and any other medications not used in the treatment of post-bariatric surgery hypoglycemia that may cause hypoglycemia or fluctuations in blood glucose levels.
  * Acetaminophen-containing products during periods of continuous glucose monitoring.

Medications such as tramadol may cause hypoglycemia or fluctuations in blood glucose levels and, as such, use of such medications is subject to the restrictions as described above during the study. Acetaminophen can interfere with the accuracy of the glucose sensor of the continuous glucose monitoring system and is, therefore, prohibited during continuous glucose monitoring.

* Major general surgery within 3 months before study entry or anticipated during the study period

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04; Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Single dose Part 1 and Multiple dose Part 2 - Incidence of treatment-emergent adverse events - | 42 days
  Safety assessed by treatment-emergent adverse events
Single dose Part 1 - Change from baseline in glucose levels | Baseline and 22 days
  Glucose measured using a continuous glucose monitor
Single dose Part 1 - Blood glucose levels | Daily through Day 11 and at Day 22
  Assessment of blood glucose with a bedside meter at multiple time points specified in the protocol
Multiple dose Part 2 - Change from baseline of duration of glucose by CGM at various levels as specified in the protocol | 28 days
  Glucose measured by continuous glucose monitoring every 5 min
Multiple dose Part 2 - Change from baseline of number of episodes and percent of episodes of hypoglycemia per day with glucose by CGM at various levels as defined in the protocol | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Allan Gordon, MD, PhD, Study Director — XOMA (US) LLC
Locations (5):
- United States (5):
  - Aurora, Colorado
  - Chicago, Illinois
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Rochester, Minnesota